CLINICAL TRIAL: NCT04391101
Title: Efficacy of Convalescent Plasma for the Treatment of Severe SARS-CoV-2 Infection: A Randomized, Open Label Clinical Trial
Brief Title: Convalescent Plasma for the Treatment of Severe SARS-CoV-2 (COVID-19)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital San Vicente Fundación (Other)
Collaborators: Clínica León XIII (Unknown); Grupo de Inmunodeficiencias primarias Universidad de Antioquia (Unknown); Clínica Universitaria Bolivariana (Unknown); Hospital Pablo Tobón Uribe (Other); Clínica Rosario El Tesoro (Unknown); Clínica Las Américas (Unknown); Clínica Cardiovid (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2020-05-08; First posted 2020-05-18 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: SARS-Cov-2
Keywords: Coronavirus; Covid-19; Convalescent plasma; Intensive Care Unit
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Open label, parallel, randomized clinical trial with stratified (center and age) patient allocation in a 2 :1 ratio (plasma: standard management) for a superiority hypothesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Administration of two units of fresh frozen plasma (between 400 and 500 ml) obtained from convalescent patients from infection by SARS-CoV-2. Convalescent plasma is defined as the plasma of patients who had PCR confirmed SARS-CoV-2 infection, who have recovered clinically, and who have positive antibodies against SARS-CoV-2.
  Interventions: Drug: Convalescent plasma
- Control group (No Intervention): Subjects assigned to the control group will receive support treatment in the intensive care unit based on institutional management guidelines. The use of antiviral, antimalarial or anti-inflammatory drugs is allowed in both groups according to the ICU protocols.

INTERVENTIONS:
Drug: Convalescent plasma — 400-500ml convalescent plasma
  Other Names: Plasma
  Arms: Intervention group

SUMMARY:
Convalescent plasma has been used for over 100 years in the treatment of severe acute respiratory infections of viral origin. There are not pharmacological treatments for the actual outbreak for SARS-Cov-2 and it is necessary to evaluate the efficacy of treatment options, including convalescent plasma transfusion. The hypothesis is that convalescent plasma is efficacious and safe for reducing mortality in patients with COVID-19 treated in ICU

DETAILED DESCRIPTION:
Coronavirus infection has been declared by the World Health Organization as a pandemic. In addition to hemodynamic and ventilatory support in the intensive care unit, there is no treatment for COVID-19. Currently proposed treatments (chloroquine, antivirals, immunomodulators, among others) have low quality studies that do not prove efficacy.

Blood or plasma transfusion from convalescent patients (patients who have overcome the disease by generating a competent immune response) has been prescribed for over 100 years. In the last 15 years, convalescent plasma has been studied for the treatment of severe acute respiratory infections of viral origin, such as severe acute respiratory syndrome (SARS), avian influenza, and influenza A (H1N1). Suppressing viremia is one of the possible explanations for the efficacy of convalescent plasma treatment.

For the treatment of COVID-19, there are case series that show a clear improvement in severe patients after administration of convalescent plasma without significant adverse events. At the current crisis of the SARS-CoV-2 pandemic, in which there are no pharmacological treatments that have proven to have any therapeutic effect, it is imperative to assess the efficacy and safety of convalescent plasma transfusion in infected patients.

This is an open, randomized clinical trial with patient allocation in a 2 :1 ratio, plasma: standard management, for a superiority hypothesis. The main objective of this study is to determine the efficacy of convalescent plasma for the treatment of severe COVID-19 infection in terms of decreased in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

For plasma donors:

* Over 18 years of age
* Men or nulliparous women with no history of recent abortions or transfusions SARS-CoV-2 infection by PCR in any sample or serological test with a maximum of 60 days from resolution of symptoms.
* If donation is done within 14 to 28 days after resolution of symptoms, the patient must have a negative PCR test for SARS-CoV-2. If donation is done after 28 days of resolving symptoms, no negative control test will be required.

For plasma recipients:

* Over 18 years of age
* SARS-CoV-2 infection confirmed by PCR in any sample
* Hospitalized in the ICU due to shock or respiratory failure, with less than 24 hours after entering the ICU.

Exclusion Criteria:

For plasma donors:

* Severe SARS-CoV-2 infections with an ICU requirement or those with asymptomatic infections will not be accepted as donors.
* Nor will a person who has received convalescent plasma as part of the COVID-19 treatment.

For plasma receivers:

* Serious volume overload or other condition that contraindicates plasma transfusion.
* History of anaphylaxis or serious adverse reaction to plasma.
* Previous diagnosis of immunoglobulin A deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Intrahospital mortality from any cause | Up to 28 days
  Proportion of patients who die while being hospitalized

SECONDARY OUTCOMES:
Length of hospital stay | Up to 60 days
  Number of days hospitalized
Free time for ventilatory support on day 60 | Day 60
  Number of days without ventilatory support
Overall survival at day 60 since hospitalization | Day 60
  Proportion of patients alive on day 60
Cumulative incidence of adverse events: transfusion reactions (fever, flare), TRALI (transfusion-associated lung injury), TACO (transfusion-related circulatory overload), transfusion- related infections | Up to 28 days
  Proportion of adverse events related with convalescent plasma

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Perilla Suarez, Hematologist, Principal Investigator — Hospital San Vicente Fundación
Locations (1):
- Hospital San Vicente Fundacion, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No